CLINICAL TRIAL: NCT02707848
Title: Epidemiological Study for Psychiatric Disorder Among Children and Adolescents
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201411056RIN
Record Dates: First submitted 2016-03-09; First posted 2016-03-14 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention

SUMMARY:
This 3-year school-based epidemiological study on child and adolescent mental disorders aims to obtain the prevalence rate and identify the psychosocial, individual, environmental, and familial risk factors for mental disorders including learning disability, autism spectrum disorder, attention-deficit hyperactivity disorder, oppositional defiant disorder, conduct disorder, mood disorders (major depression, dysthymia, bipolar disorder), anxiety disorders, phobia, obsessive compulsive disorder, sleep disorders, eating disorders, and substance use disorders in Taiwan.

DETAILED DESCRIPTION:
Despite several waves of epidemiological studies in adult and elderly mental disorders in the past decades, revealing inconsistent results, little is known about the prevalence of mental disorders in the child and young adolescent population in Taiwan. However, there is an increasing trend of child and adolescent mental disorders over the past decades consistently reported across countries. With the revision of the Diagnostic and Statistical Manual of Mental Disorders to the current version-5th edition (DSM-5), there has been no epidemiological study using DSM-5 in youth population in the world. The DSM-5 was published in October 2014. It warrants an epidemiological study on child and adolescent mental disorders using the DSM-5 as diagnostic criteria in Taiwan.

This is a two-stage design to conduct screening for mental disorders including autism and all neuropsychological studies in addition to questionnaires. Moreover, clinical assessment will be conducted among urban students (n = 3000) and rural students (n = 1500) from a three-stage cluster sampling. All the screen positive (estimated n = 900) and 10% of screen negative (estimated n = 360) will receive the full diagnostic interview (K-SADS-E to obtain the pregnancy, developmental and medical history. For students who leave of absence, we will visit them at home to complete all the assessments.

The investigators anticipate this study will provide the prevalence of a wide range of developmental and psychiatric disorders in children and our results will also provide a comprehensive risk factors for each psychiatric disorder identified in this study, including neurocognitive, developmental, familiar, and environmental factors. The individual, combined, and interactive effects of these predictors can be identified in this study. This study will definitely provide precious data for the government to develop a preventive program for mental disorders and a promotion program for mental health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* urban students (n = 3000) and rural students (n = 1500) from a three-stage cluster sampling

Exclusion Criteria:

-

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: School students aged 8-14 in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Screening for mental disorders | 2 hours
  Schedule for affective disorders and schizophrenia for school-age children revision (K-SADS-E), Autism Diagnostic Observation Schedule (ADOS)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lin HT, Tai YM, Gau SS. Autistic Traits and Cyberbullying Involvement Mediated by Psychopathologies and School Functions in a Nationally Representative Child Sample. Cyberpsychol Behav Soc Netw. 2023 Sep;26(9):706-716. doi: 10.1089/cyber.2022.0309. Epub 2023 Jul 21. PMID 37477877